CLINICAL TRIAL: NCT04217382
Title: Pre Transplantation Melanoma : Retrospective and Prospective Multicenter Observational Study
Brief Title: Pre Transplantation Melanoma
Acronym: MPG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0636
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient with melanoma pre transplantation — survival time without melanoma recurrence

SUMMARY:
Melanoma incidence is increase in global population and number of transplantation also. However immunosuppressor increase recurrence risk of melanoma.

There are more and more cases of eligible patients to transplant with an antecedent of melanoma. There is no guideline yet.

Main objective is survival time without melanoma recurrence in this population to do guideline of time limit or not between melanoma and transplantation by stage.

ELIGIBILITY:
Inclusion Criteria:

* patient with an antecedent of melanoma before transplantation
* Not opposite to participate

Exclusion Criteria:

* Under the age of 18
* patient under Guardianship
* patient not affiliated with a health system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with an antecedent of melanoma before transplantation
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
survival time without melanoma recurrence | at enrollment
  Delay in recurrence-free survival since diagnosis and since transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Emilie DUCROUX, MD, Principal Investigator — Service de Dermatologie, Hôpital Edouard Herriot, Lyon
Locations (1):
- service de dermatologie - hopital Edouard Herriot, Lyon, Rhone, France